CLINICAL TRIAL: NCT00850837
Title: Safety of Acidform Lubricant (Amphora) in Women at Low Risk for HIV-1 Infection
Brief Title: Safety of Acidform Lubricant in HIV-Uninfected Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Keller 069551 AF020; U01AI069551 (NIH); 10740 (Registry Identifier: DAIDS ES); AF 020
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: Microbicide; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will apply Acidform lubricant twice daily for 14 consecutive days between menses
  Interventions: Drug: Acidform Lubricant
- 2 (Placebo Comparator): Participants will apply HEC gel twice daily for 14 consecutive days between menses
  Interventions: Drug: HEC gel

INTERVENTIONS:
Drug: Acidform Lubricant — 5 g application of acid buffered gel (pH = 3.5)
  Other Names: Amphora
  Arms: 1
Drug: HEC gel — 5 g application of hydroxyethylcellulose gel
  Arms: 2

SUMMARY:
Topical microbicides, substances that kill microbes, are being studied to prevent sexual transmission of HIV and other disease pathogens. In the future, topical microbicides may be applied vaginally to prevent both acquisition and transmission of HIV and other sexually transmitted infections (STIs). The purpose of this study is to compare the safety of daily applications of Acidform lubricant and HEC gel in healthy women at low risk for HIV infection and assess the effect of a microbicide candidate on the natural immunity women have to STI pathogens.

DETAILED DESCRIPTION:
A new approach to HIV prevention currently being studied is the use of topical microbicides. This study will measure the mucosal response to daily intravaginal applications of Acidform lubricant and HEC gel in two groups of healthy women at low risk for HIV infection.

The duration of this study for each participant is 3 weeks. Study participants will be randomly assigned to one of two study groups. Group 1 participants will apply Acidform lubricant twice daily for 14 consecutive days between menses. Group 2 participants will apply HEC gel for 14 consecutive days between menses.

After screening and study entry, study visits will occur on Days 7, 14, and 21. Study entry will occur 2 to 6 days following the menses and within 45 days of screening. Medical and sexual history, a pelvic exam, cervicovaginal lavage sample collection, blood collection, vaginal pH testing, STI testing, and adverse effect reporting will occur at all visits. Cytobrush collection, vaginal swab, and cervical biopsy will occur at selected visits. All participants will be asked to complete a diary throughout the study; this diary will be reviewed at all study visits. A Pap smear will be obtained at screening if documentation of a negative Pap smear result within the last year is not available.

ELIGIBILITY:
Inclusion Criteria:

* Normal menstrual history with regular cycles and with a minimum of 21 days between menses
* Low risk for HIV/STI infection. More information on this criterion can be found in the protocol.
* Agree to abstain from vaginal and anal intercourse and to not use vaginal products within 48 hours prior to study entry and for the duration of the study

Exclusion Criteria:

* HIV-infected
* Menopausal
* Currently using hormonal contraception or have used hormonal contraception within 2 months of study entry
* Menstruating at screening or enrollment visits
* Urinary tract infection at screening
* Positive chlamydia, gonorrhea, or trichomonas result at screening
* Abnormal Pap smear
* Clinically detectable genital abnormality. More information on this criterion can be found in the protocol.
* Currently participating in a research study of other vaginal products
* History of intermenstrual bleeding within 3 months prior to study entry
* Previous gynecologic surgery or have received treatment for syphilis, genital herpes, chlamydia, gonorrhea, trichomonas, or genital warts within 6 months prior to study entry
* Received treatment for Candida, bacterial vaginosis, or urinary tract infection within 1 month prior to study entry
* Have douched or used vaginal products, including lubricants, feminine hygiene products, vaginal drying agents, and sex toys within 48 hours prior to study entry
* Vaginal or anal intercourse during the 48 hours prior to study entry
* Oral antibiotics within 7 days of study entry
* Pregnant, less than 6 months postpartum, or breastfeeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2009-02

PRIMARY OUTCOMES:
Measured endogenous antimicrobial activity | Throughout study
Measured levels of mediators of host defense, including defensins, cytokines, and chemokines in CVL | Throughout study

SECONDARY OUTCOMES:
Extent and duration of buffering measured by vaginal pH | Prior to and 2 hours after first application
Changes in epithelial integrity after Acidform and HEC application | Throughout study
Changes in vaginal flora following Acidform and HEC application | Throughout study
Antiviral activity in CVL following Acidform and HEC application | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Marla Keller, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine - East Campus GCRC (Herold) Non-Network CRS, The Bronx, New York, United States

REFERENCES:
- [Background] Anderson DJ, Williams DL, Ballagh SA, Barnhart K, Creinin MD, Newman DR, Bowman FP, Politch JA, Duerr AC, Jamieson DJ. Safety analysis of the diaphragm in combination with lubricant or acidifying microbicide gels: effects on markers of inflammation and innate immunity in cervicovaginal fluid. Am J Reprod Immunol. 2009 Feb;61(2):121-9. doi: 10.1111/j.1600-0897.2008.00670.x. PMID 19143675
- [Background] Behets FM, Turner AN, Van Damme K, Rabenja NL, Ravelomanana N, Swezey TA, Bell AJ, Newman DR, Williams DL, Jamieson DJ; Mad STI Prevention Group. Vaginal microbicide and diaphragm use for sexually transmitted infection prevention: a randomized acceptability and feasibility study among high-risk women in Madagascar. Sex Transm Dis. 2008 Sep;35(9):818-26. doi: 10.1097/OLQ.0b013e318175d8ab. PMID 18562985
- [Background] Williams DL, Newman DR, Ballagh SA, Creinin MD, Barnhart K, Weiner DH, Bell AJ, Jamieson DJ. Phase I safety trial of two vaginal microbicide gels (Acidform or BufferGel) used with a diaphragm compared to KY jelly used with a diaphragm. Sex Transm Dis. 2007 Dec;34(12):977-84. doi: 10.1097/olq.0b013e31813347e9. PMID 18080349
- [Derived] Keller MJ, Carpenter CA, Lo Y, Einstein MH, Liu C, Fredricks DN, Herold BC. Phase I randomized safety study of twice daily dosing of acidform vaginal gel: candidate antimicrobial contraceptive. PLoS One. 2012;7(10):e46901. doi: 10.1371/journal.pone.0046901. Epub 2012 Oct 8. PMID 23056520